CLINICAL TRIAL: NCT03235206
Title: Massage Therapy and the Well-Being of Police Officers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alanah Whiteway (Other)
Responsible Party: Sponsor-Investigator, Alanah Whiteway, Student, Academy Canada
Organization: Academy Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTPO
Record Dates: First submitted 2017-07-24; First posted 2017-08-01 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Occupational Problems; Occupational Injuries; Occupation-related Stress Disorder
Keywords: Police Officers
MeSH Terms: conditions — Occupational Injuries | interventions — Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Massage Therapy — This study will compare surveys taken before the participants began their massage treatments, and after 12 one hour massages. These surveys will judge sleep quality, stress levels, and mental health during varying days in the participants work cycle. It will also compare a postural assessment and range of motion testing done before the first treatment and after the last.

SUMMARY:
This study is intend to show the positive impact that massage therapy can have on the lives of police officers. The study will demonstrate how regular treatment can change sleeping quality, stress levels and mental health. It will also investigate the impact that police work can have on the body.

ELIGIBILITY:
Inclusion Criteria:

* Police Officers preferable working on the street within the St. John's area

Exclusion Criteria:

* Civilians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Muscular Imbalances | After 12 one hour massages
  A measure of any muscular imbalances that present in each clients. All client findings will be compared to see if there is a pattern through the participants. Clients will have notes compared from the beginning to the end as well to see if there has been any improvement.
Postural Dysfunctions | After 12 one hour massages
  A postural assessment will be done at the beginning of the study and then be compared to one done at the end to see if there have been any improvements. All clients postural assessments will be compared to see if there is any pattern among participants. The main focus will be on the back and hip.
Range of Motion | After 12 one hour massages
  The range of motion of major joints will be assess to see if they fall within the norm, or if each client is limited. The client will have a range of motion test done at the beginning of treatment and again at the end to see if there has been any improvement. All clients range of motion testing will be compared to see if there are any patterns throughout the officers.

SECONDARY OUTCOMES:
Stress Levels | After 12 one hour massages
  Stress levels will be rated on a scale of 1 to 5 (one being no stress and 5 being extremely stressed) to see if during the duration of the study they find a decrease in their stress levels.
Sleep Quality | After 12 one hour massages
  To see if there is improvement of sleep quality in general, and sleep quality during change over shifts. Sleep will be rated on a scale of 1 to 5 (One being no sleep and five being a complete night of uninterrupted sleep). This will compared from studies completed throughout the study.
Mental Wellness | After 12 one hour massages
  The clients will be asked to fill out a survey throughout the study on how the feel mental. It will be rated on a scale of 1 to 5 (one be extremely depressed and 5 being over the moon happy) These will be compared from the beginning to the end of treatment to see if there is any improvements.

IPD SHARING:
Plan to Share IPD: Undecided